CLINICAL TRIAL: NCT04226508
Title: Different Modalities of Exercise for Physical Activity Promotion in Cancer Patients
Brief Title: "CHOiCE"! Choose Health: Oncological Patients Cenetered Exercise
Acronym: CHOiCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Alice Avancini, Investigator, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 33320
Record Dates: First submitted 2019-12-20; First posted 2020-01-13 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Mixed Cancer
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The CHOiCE includes different substudies, with different study designs, i.e., RCT, single arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Physical exercise (Experimental)
  Interventions: Other: Physical exercise

INTERVENTIONS:
Other: Physical exercise — The patients can choose between three modality of EX:
  1. Autonomous supervised training : a personalized activity is proposed. People choosing this modality have a written material, in which all the exercise, the activity, the frequency, the duration, the intensity are specifically described and reported, to perform the training at home. A training diary and 7 meetings (face to face, or skype or other modality) are proposed for monitoring the intervention.
  2. Personal training program: a personalized activity is proposed. Patients are followed individually in a gym contest by a qualified kinesiologist.
  3. Group training program: the training is performed in a small group, supervised and monitored by a qualified kinesiologist. The instructor-user ratio is 1:4 - 1:8, depending on the functional conditions and the heterogeneity of the participants.
  Arms: Physical exercise

SUMMARY:
The "CHOICE!" study is an exercise program following the recommendation of the American College of Sports Science for cancer patients. The aims of the intervention are to test the safety and feasibility of a structured program, letting patients choose the modality of delivery. Secondary endpoints include exercise health-related skills and quality of life. The program considers the preferences of exercise of cancer survivors, giving the possibility to choose the exercise modality (autonomous, with a personal trainer or group class). This program will be tested in different cancer populations with different study designs based on different patients cohort (i.e., RCT or single-arm).

ELIGIBILITY:
Inclusion Criteria:

* a confirmed cancer diagnosis;
* ≥ 8 weeks post-surgical procedure;
* Medical clearance for participation provided by primary care physician or oncologist;
* Informed consent signed;

Exclusion Criteria:

* Age < 18 years old;
* Pregnancy;
* Inability to ambulate;
* Contraindication to participation in a regular physical activity program;
* Inability to understand the instructions for PA and/or Mini Mental State index <24;
* Serious physical limitation and/or Karnofsky index <50.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
The number of participants with an adverse event | Change from baseline to 12 weeks
  Adverse events will categorize according to the Common Terminology Criteria for Adverse Events (version 5.0)
The eligibility rate | At 12 weeks
  The number of patients considered eligible dividing the number of subjects who meet inclusion criteria
The recruitment rate | At 12 weeks
  The number of patients randomized dividing the number of subjects considered eligible
The adherence to exercise protocol | At 12 weeks
  Measured by the total number of exercise sessions attended
The dropouts rate | At 6 months
  Defined as a participant who leaves the study for any reason prior to completing the 12-week (24 session) exercise program. All reasons for drop out will be reported.

SECONDARY OUTCOMES:
Cardiorespiratory fitness | Change from baseline cardiorespiratory fitness at 3 months
  Using the Six minutes walking test
Upper limb muscle strength | Change from baseline muscle strength at 3 months
  Using the Handgrip strength test
Lower limb muscle strength | Change from baseline muscle strength at 3 months
  Using the Isometric Leg Press strength test
Upper limb flexibility | Change from baseline flexibility at 3 months
  Using the Back Scratch test
Lower limb flexibility | Change from baseline flexibility at 3 months
  Using the Sit and Reach test
Body mass index | Change from baseline antrhopometric values at 3 months
  Calculated from weight and height
Waist-hip ratio | Change from baseline antrhopometric values at 3 months
  Calculated usign the waist and hip circumferences
Enjoyment | Change from baseline enjoyment at 3 months
  Using the Physical Activity Enjoyment Scale (PACES), ranging from 0 (no enjoyment) to 75 (max enjoyment)
Quality of life (QoL) | Change from baseline quality of life at 3 months
  Using European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ C-30), ranging from 0 (lowest QoL) to 100 (highest QoL)
Physical activity level | Change from baseline physical activity level at 3 months
  Using the Godin's Leisure Time Exercise Questionnaire (GLTEQ). GLTEQ inquires about frequency of vigorous, moderate and mild intensity EX as defined by Godin. Subsequently, each frequency is multiplied by its correspondent metabolic equivalent of the task (MET), i.e. vigorous*9; moderate*5; mild*3. A Leisure Score Index (LSI) was calculated, using the sum of vigorous and moderate components. Based on LSI patients were then classified as active (if LSI≥ 24) and insufficiently active (if LSI<24) according to the American College of Sport Medicine Physical Activity Guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Lanza, Principal Investigator — Universita di Verona
Locations (2):
- Italy (2):
  - Italian League for Fight Cancer, Biella, Turin
  - University of Verona, Verona

REFERENCES:
- [Derived] Avancini A, Borsati A, Baldo E, Ciurnelli C, Trestini I, Tregnago D, Belluomini L, Sposito M, Insolda J, Auriemma A, Fiorio E, Piacentini M, Schena F, Milella M, Pilotto S. A Feasibility Study Investigating an Exercise Program in Metastatic Cancer Based on the Patient-Preferred Delivery Mode. Oncologist. 2024 Jun 3;29(6):e828-e836. doi: 10.1093/oncolo/oyae002. PMID 38206849